CLINICAL TRIAL: NCT05260073
Title: A Prospective Cohort Study of Patients With Actinic Keratosis (AK) in the Face or Scalp Treated With Tirbanibulin and Followed for 24 Weeks Post Treatment-initiation. Patient Reported Outcomes (PROs) and Clinical Profile of Patients Will be Gathered for Descriptive Analyses of Patient Outcomes Over the 24-week Study Observation Period
Brief Title: Patient and Clinician Reported Outcomes for Tirbanibulin Effectiveness and Safety in Actinic Keratosis
Acronym: PROAK
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: M-14789-43
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic | interventions — tirbanibulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tirbanibulin: Participants will receive tirbanibulin ointment 2.5 mg in 250 mg (single dose packet). The participants will be observed for 24 weeks to gather participant reported outcomes (PROs) and clinical profile.
  Interventions: Drug: Tirbanibulin

INTERVENTIONS:
Drug: Tirbanibulin — Participants will be treated with tirbanibulin ointment 1% (2.5 mg tirbanibulin in 250 mg) as 1 single-dose packet per application, for 5 consecutive days.
  Other Names: Klisyri®

SUMMARY:
The purpose of the study is to evaluate patient reported outcomes (PROs) in terms of health-related quality of life (HRQoL) among subjects with actinic keratosis (AK).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AK of the face or scalp
* Has clinically typical, visible, and discrete AK lesions
* Considered as a potential candidate for tirbanibulin (Klisyri®) treatment to manage their AK
* Willing to avoid excessive sun or ultraviolet (UV) exposure, and/or use relevant sunscreen protection and protective clothing during the study duration
* Able to read and write English
* Provide consent to participate in the study
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Participants with any dermatological condition of the face or scalp that could interfere with the clinical evaluations.
* Hypertrophic AK lesions, open wounds or suspected skin cancers within close proximity of the treatment area.
* Anticipated need for in-patient hospitalization or in-patient surgery within the next 2 months.
* Participants unable to comply with the requirements of the study or participants who in the opinion of the study physician should not participate in the study.
* Participants for whom medical chart is inaccessible to physicians to complete baseline data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be participants diagnosed with AK on the face or scalp, and aged 18 years or above at the time of initiation of treatment. The study cohort will be drawn from dermatology clinics from across the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Almirall Investigational Site 1, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berman B, Armstrong A, Lebwohl M, Grada A, Bhatia N, Patel VA, Rigel D, Del Rosso J, Schlesinger T, Kircik L, Salem R, Narayanan S, Kasujee I. Developing a questionnaire for assessing clinician- and patient-reported outcomes in actinic keratosis: Results from an expert panel. JAAD Int. 2023 Sep 23;16:192-198. doi: 10.1016/j.jdin.2023.09.006. eCollection 2024 Sep. PMID 39040844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 32 sites in the United States from 9 March 2022 to 7 March 2023.
Pre-assignment Details: A total of 300 participants were enrolled, out of which 290 participants who completed the week 8 study survey were included in the full analysis set.
Groups:
- Tirbanibulin: Participants with actinic keratosis (AK) applied tirbanibulin ointment 1% topically once daily using 1 single-dose packet (2.5 milligrams [mg] in 250 mg) per application, for 5 consecutive days were observed for 24 weeks to gather participant reported outcomes (PROs) and clinical profile.
Period: Overall Study
Arm/Group | Tirbanibulin
Started | 300
Full Analysis Set (Full Analysis Set (FAS) included all participants who received at least one dose of tirbanibulin during the study observation period of 8-weeks related to primary endpoint, as part of usual care and had at least some data pertaining to the key variables studied at relevant timepoints, post-baseline.) | 290
Completed | 279
Not Completed | 21
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Population: FAS included all participants who received at least one dose of tirbanibulin during the study observation period of 8-weeks related to primary endpoint, as part of usual care and had at least some data pertaining to the key variables studied at relevant timepoints, post-baseline.
Groups:
- Tirbanibulin: Participants with AK applied tirbanibulin ointment 1% topically once daily using 1 single-dose packet (2.5 mg in 250 mg) per application, for 5 consecutive days were observed for 24 weeks to gather PROs and clinical profile.
Arm/Group | Tirbanibulin
Number analyzed (Participants) | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.30 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 269
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 285
  Race: Black or African American | 0
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Other | 2
  Race: Prefer not to answer | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Domain Scores Using the Patient Reported Outcome Skindex-16 Instrument at Week 8
Description: Skindex-16 is a validated dermatological instrument to measure dermatology-specific Health-Related Quality of Life (HRQoL). The Skindex-16 consisted of 16 items that were divided into three domains: Symptoms (four items, range 0-24), Emotions (seven items, range 0-42), and Functioning (five items, range 0-30). Participant were asked to respond on how much their skin condition bothered them in the week prior to administration of the Skindex-16. Each item was scored on a scale ranged from 0 (never bothered) to 6 (always bothered), where higher score indicated continued/more botheration. Item scores are transformed to 0 to 100 scale, and domain scores are calculated as the average of the item scores comprising the domain. Net positive changes in respective subscale scoring indicates improvement in that particular Quality of life assessment (i.e., Symptoms, Emotions, Functioning), while net negative changes in scoring indicates decrease in that particular Quality of life assessment.
Time Frame: Baseline, Week 8
Population: FAS included all participants who received at least one dose of tirbanibulin during the study observation period of 8-weeks related to primary endpoint, as part of usual care and had at least some data pertaining to the key variables studied at relevant timepoints, post-baseline. Here, "number analyzed" signifies participants who were evaluable at each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tirbanibulin
Number analyzed (Participants) | 290
score on a scale
  Symptoms Domain Score: Baseline: number analyzed (Participants) | 289
  Symptoms Domain Score: Baseline | 22.30 (22.36)
  Symptoms Domain Score: Change at Week 8: number analyzed (Participants) | 289
  Symptoms Domain Score: Change at Week 8 | -14.26 (27.77)
  Emotions Domain Score: Baseline: number analyzed (Participants) | 286
  Emotions Domain Score: Baseline | 38.17 (27.30)
  Emotions Domain Score: Change at Week 8: number analyzed (Participants) | 286
  Emotions Domain Score: Change at Week 8 | -24.88 (32.96)
  Functioning Domain Score: Baseline | 14.41 (20.06)
  Functioning Domain Score: Change at Week 8 | -9.78 (23.66)

2. Secondary Outcome: Percentage of Participants With Investigator Global Assement (IGA) Success at Week 8
Description: IGA success was defined as achieving a rating of 'completely cleared' (0) or 'partially cleared' (1) in IGA of AK status at Week 8. The IGA is 5-point scale that assessed the severity of actinic keratosis, with scores ranged from 0 (completely clear) to 4 (not cleared): 0 = completely cleared (100% clearance); 1 = partially cleared (>=75% clearance); 2 = moderately cleared (50% to 74% clearance); 3 = minimally cleared (<50% clearance); 4 = not cleared (0% clearance), where higher score indicated higher severity.
Time Frame: At Week 8
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tirbanibulin
Number analyzed (Participants) | 290
percentage of participants | 73.79

ADVERSE EVENTS:
Time Frame: From start of study up to end of the study (Week 24)
Description: Safety population included all participants who received at least one dose of tirbanibulin during the study observation period of 8-weeks related to primary endpoint, as part of usual care.
Arm/Group | Tirbanibulin
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 6/300
Other Adverse Events (participants affected / at risk) | 9/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirbanibulin (N=300)
Fall (Injury, poisoning and procedural complications) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirbanibulin (N=300)
COVID-19 (Infections and infestations) | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Capillary fragility (Vascular disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT05260073/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT05260073/SAP_001.pdf